CLINICAL TRIAL: NCT01057550
Title: A Randomised Controlled Trial Comparing TVT, Pelvicol and Autologous Fascial Slings for the Treatment of Stress Urinary Incontinence in Women
Brief Title: Randomised Controlled Trial Comparing Tension-Free Vaginal Tape (TVT), Pelvicol & Autologous Slings for Stress Urinary Incontinence(SUI)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abertawe Bro Morgannwg University NHS Trust (Other Government)
Collaborators: C. R. Bard (Industry)
Responsible Party: Dr Karen Guerrero, ABM University Hospital NHS Trust
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2000.117
Record Dates: First submitted 2010-01-26; First posted 2010-01-27 (Estimated); Last update posted 2010-01-27 (Estimated); Status verified 2004-03

CONDITIONS: Stress Urinary Incontinence
Keywords: Stress urinary Incontinence; autologous slings; slings; tvt; grafts; surgery
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Autologous Fascial Sling (Active Comparator): Retropubic, bottom up autologous sling
  Interventions: Procedure: Autologous fascial sling
- TVT (Active Comparator): Standard retropubic TVT
  Interventions: Procedure: TVT
- Pelvicol (Active Comparator): Retropubic mid urethral sling made from Pelvicol
  Interventions: Procedure: Pelvicol

INTERVENTIONS:
Procedure: Autologous fascial sling — Retropubic bottom up mid urethral sling made using autologous rectus sheath fascia
  Arms: Autologous Fascial Sling
Procedure: TVT — Standard TVT as described by Ulmsten 1996
  Arms: TVT
Procedure: Pelvicol — retropubic mid urethral sling made from Pelvicol
  Arms: Pelvicol

SUMMARY:
The purpose of this trial was to discover which type of operation for stress urinary incontinence in women offered better results: autologous slings, TVT or Pelvicol slings.

ELIGIBILITY:
Inclusion Criteria:

* Women requiring surgery for SUI following failed conservative treatment

Exclusion Criteria:

* Under 18 years of age
* Previous surgery for SUI
* Evidence of neurological disease
* Pelvic Organ Prolapse (POP) greater than Grade 2
* Women with any evidence of Detrusor Overactivity or bladder hypocompliance on urodynamic assessment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2001-10; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
success rate at improving symptom of stress urinary incontinence | 1 year

SECONDARY OUTCOMES:
completely dry rates | 1 year
quality of life scores | 1 year
intra & post-operative complications | 1 year
re-operation rates | 1 year
hospital stay | 5 days
operative time | hours

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm G Lucas, Study Chair — ABM University Hospital NHS trust
Locations (1):
- ABM University Hospital NHS trust, Swansea, Wales, United Kingdom

REFERENCES:
- [Result] Guerrero KL, Emery SJ, Wareham K, Ismail S, Watkins A, Lucas MG. A randomised controlled trial comparing TVT, Pelvicol and autologous fascial slings for the treatment of stress urinary incontinence in women. BJOG. 2010 Nov;117(12):1493-502. doi: 10.1111/j.1471-0528.2010.02696.x. Epub 2010 Sep 24. PMID 20939862